CLINICAL TRIAL: NCT04689516
Title: The Use of Thoracic Fluid Content as a Guide for 6% HES Infusion During Hypervolemic Hemodilution in Patients With Placenta Accreta. A Randomized Controlled Trial.
Brief Title: Thoracic Fluid Content During Hypervolemic Hemodilution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherif Abdullah Mohamed, Lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: N- 25 / 2020
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Edema
Keywords: Thoracic fluid content; lung ultrasound; cesarean section; placenta accreta; colloid
MeSH Terms: conditions — Pulmonary Edema; Placenta Accreta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): will receive a hypervolemic hemodilution with an IV infusion load of 6% HES.The infusion will be started preoperatively and will stop after completion of the infused volume. LUS evaluation will be done before start and after the end of the infusion.
  Interventions: Device: Thoracic fluid content estimation
- The TFC Group (Experimental): will receive hypervolemic hemodilution with an IV infusion load of 6% HES.The infusion will be started preoperatively . The patient will be monitored for thoracic fluid content and LUS score. The infusion will stop if TFC reaches 40 k ohm-1 or after completion of the infused volume. LUS evaluation will be done before start and after the end of the infusion.
  Interventions: Device: Thoracic fluid content estimation

INTERVENTIONS:
Device: Thoracic fluid content estimation — The patient will be monitored for thoracic fluid content and LUS score. The infusion will stop if TFC reaches 40 k ohm-1 or after completion of the infused volume. LUS evaluation will be done before the start and after the end of the infusion.
  Other Names: extravascular lung water estimation

SUMMARY:
Thoracic fluid content (TFC) is one of the many variables measured by the ICON electrical cardiometry (EC) device (Osypka Medical). The ICON device is often called "thoracic electrical bio-impedance" that based on measuring the changes in total resistance of the thorax to electric current and is considered a numerical measure of total (intravascular and extravascular) thoracic fluid. Although TFC is a measure of both extra and intra-vascular thoracic fluid, it provides an estimate of the increase in intrathoracic fluids such as to facilitate the risk of pulmonary edema.

Although many studies were done on the ability of TFC to detect pulmonary edema in preeclampsia, ARDS, heart failure, weaning from mechanical ventilation and during fluid management in prolonged surgery , yet, there is no study before was done on the use of TFC as a guide for fluid therapy during hypervolemic hemodilution in major obstetric surgery in patients with placenta accreta as one of the most common etiologies of life-threatening obstetric hemorrhage and the most common cause of peripartum hysterectomy

Aim of the work:

To use TFC as a guide for 6% HES infusion of hypervolemic hemodilution in patients with placenta accreta to avoid fluid overload.

Objectives:

* To calculate LUS score at the end of infusion.
* To evaluate TFC in k ohm-1.
* To assess oxygen saturation, PO2 and P/F ratio in ABG.
* To calculate the total infused volume in milliliters.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18-45 years old
* ASA I-II

Exclusion Criteria:

* younger than 18 years,
* ASA > or = III
* patients with respiratory, cardiac disease, cardiac arrhythmias,
* body mass index above 40 kg/m2
* renal insufficiency,
* sepsis,
* hypovolemia denoted by PPV > 13 detected after start of mechanical ventilation,
* preoperative baseline LUS score 10 or more,
* TFC > or = 26 k ohm-1,
* patients with neck or chest lesions that impair the application of cardiometry electrodes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cesarean section patients
Enrollment: 56 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
detection of pulmonary edema | 30 minutes after start infusion
  thoracic fluid content estimation using cardiometry and lung ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University hospitals, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] Spahn DR, Theusinger OM, Hofmann A. Patient blood management is a win-win: a wake-up call. Br J Anaesth. 2012 Jun;108(6):889-92. doi: 10.1093/bja/aes166. No abstract available. PMID 22593125
- [Background] Kunst PW, Vonk Noordegraaf A, Raaijmakers E, Bakker J, Groeneveld AB, Postmus PE, de Vries PM. Electrical impedance tomography in the assessment of extravascular lung water in noncardiogenic acute respiratory failure. Chest. 1999 Dec;116(6):1695-702. doi: 10.1378/chest.116.6.1695. PMID 10593797
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031